CLINICAL TRIAL: NCT02813213
Title: Effectiveness Comparison Between the Use of Skin Micro-grafts vs Meshed Split Thickness Skin Grafts in Cutaneous Defects: A Randomized Controlled Clinical Trial
Brief Title: Effectiveness Comparison of Skin Micro-grafts vs Meshed Split Thickness Skin Grafts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Alejandro Cruz Segura, MD, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2013-3501-8
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Skin Ulcer; Burns
Keywords: skin transplantation; grafting skin
MeSH Terms: conditions — Skin Ulcer; Burns | interventions — Skin Transplantation

STUDY DESIGN:
Intervention Model Description: Experimental intervention: skin micro grafts Comparative intervention: Meshed Split Thikness Skin Grafts
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard skin graft (Active Comparator): This group is comprised of patients' wound halves that will receive meshed (1:3) split thickness skin graft (0.3-0.5mm thickness). This half will be covered with a standard "tie over" dressing. The dressing will be removed at day 5, and then it will be removed every 3 days up to the 14th day.
  Interventions: Procedure: Standard skin graft
- Skin micro graft (Experimental): This group is comprised of the patients' wound halves that will receive skin micro grafts. To obtain this grafts the investigators will use "Xpansion micro-autografting" system. They will use 0.8 x 0.8 mm skin grafts with a graft to graft distance of 4mm (1:50 expansion).This half will be covered with a special hydrogel dressing with keratinocyte growth factor (Epilife medium with calcium) 1.5ml for each 14 square centimeters of the wound. This half will be covered with a wet adhesive foam dressing and then it will be covered up with a non-adherent interface dressing (tegaderm). The dressing will be removed at day 5, and then it will be removed every 3 days up to the 14th day. Each time of dressing change only the non-adherent interface dressing will be removed, and the area will be bathed with keratinocyte growth factor solution.
  Interventions: Procedure: Skin micro Grafts

INTERVENTIONS:
Procedure: Skin micro Grafts — 0.8 x 0.8 skin micro graft with graft to graft distance of 4 cm (1:50 expansion) bathed with keratinocyte growth factor solution ( 1.5 ml for each 14 square centimeters of wound)
  Other Names: Xpansion micro auto grafting system; micro grafts
  Arms: Skin micro graft
Procedure: Standard skin graft — Standard split thickness (0.3-0.5mm) skin graft
  Other Names: split thickness skin graft; skin grafting; skin grafts; medium split thickness skin graft
  Arms: Standard skin graft

SUMMARY:
This is a double-blind randomized controlled clinical trial, that compares the percentage of epithelialization of skin defects using the conventional meshed split thickness skin grafts vs skin micro grafts.

Two techniques will be applied in the same patient. The skin defect will be divided in two parts, and with a randomized method each half of this defect will be assigned to one of the two techniques.

DETAILED DESCRIPTION:
Split thickness skin graft is the standard technique in skin defects reconstruction.

The etiology of this problem is diverse (burns, infections, trauma, cancer) however, many times the availability of donor areas are insufficient and morbidity and complications that may arise make prohibitive the use of this technique in many situations.

Skin micro grafts technique consists in using a very small part of skin (0.8x 0.8 mm) and keratinocyte growth-factor solution that allows a 1:50- 1:100 skin expansion. It has many advantages: it can be performed with local anesthesia and donor area is tiny.

The study consists in using the conventional and the new technique in the same patient. The skin defect will be divided in two parts, and with a randomized method each half of this defect will be assigned to one of the two different techniques. The result variable will be the "percentage of epithelialization" and will be compared in the two halves. This variable will be measured at day 14 using clinical and image software methods. The patient and the investigator that record the outcome variable will be blinded to the type of technique.

The investigators will take skin biopsies of two halves and will perform pathology studies.

ELIGIBILITY:
Inclusion Criteria:

* Non complicated wounds (no infection, no cancer)
* Wound area: 20 x 20 cms or less
* Located in diverse anatomical regions (except axillar, groin, genital, sole, scalp and flexion or extension areas)

Exclusion Criteria:

* High cardiovascular risk
* Patients with indication of a different technique

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of epithelialization | 14th day
  It will be measured with imaging software (comparing color density) in order to calculate the percentage of epithelialization at day 14 compared with the initial wound area

SECONDARY OUTCOMES:
Histological study | 14th day
  Study of the histological characteristics of the skin under microscope
Clinical percentage of epithelialization | 14th day
  It will be measured with the "irregular patterns" technique that uses different sizes of geometric patterns in order to calculate the area of a irregular surface. Epithelialization will be compared at day 14 compared with the initial wound area.

CONTACTS AND LOCATIONS:
Locations (1):
- "La Raza" Medical Center. IMSS, Azcapotzalco, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Only some data will be shared (age, gender, diagnosis, area defect and epithelialization ratio). Photos will be shared only if the patients give their consent.

REFERENCES:
- [Result] Chern PL, Baum CL, Arpey CJ. Biologic dressings: current applications and limitations in dermatologic surgery. Dermatol Surg. 2009 Jun;35(6):891-906. doi: 10.1111/j.1524-4725.2009.01153.x. Epub 2009 Apr 6. PMID 19397669
- [Result] MEEK CP. Successful microdermagrafting using the Meek-Wall microdermatome. Am J Surg. 1958 Oct;96(4):557-8. doi: 10.1016/0002-9610(58)90975-9. No abstract available. PMID 13571547
- [Result] MEEK CP. Extensive severe burn treated with enzymatic debridement and microdermagrafting: case report. Am Surg. 1963 Jan;29:61-4. No abstract available. PMID 13934413
- [Result] TANNER JC Jr, VANDEPUT J, OLLEY JF. THE MESH SKIN GRAFT. Plast Reconstr Surg. 1964 Sep;34:287-92. No abstract available. PMID 14209177
- [Result] Green H, Rheinwald JG, Sun TT. Properties of an epithelial cell type in culture: the epidermal keratinocyte and its dependence on products of the fibroblast. Prog Clin Biol Res. 1977;17:493-500. PMID 928463
- [Result] Rheinwald JG, Green H. Serial cultivation of strains of human epidermal keratinocytes: the formation of keratinizing colonies from single cells. Cell. 1975 Nov;6(3):331-43. doi: 10.1016/s0092-8674(75)80001-8. PMID 1052771
- [Result] Munster AM. Use of cultured epidermal autograft in ten patients. J Burn Care Rehabil. 1992 Jan-Feb;13(1):124-6. doi: 10.1097/00004630-199201000-00028. PMID 1572841
- [Result] Wood FM, Stoner M. Implication of basement membrane development on the underlying scar in partial-thickness burn injury. Burns. 1996 Sep;22(6):459-62. doi: 10.1016/0305-4179(95)00178-6. PMID 8884006
- [Result] Chester DL, Balderson DS, Papini RP. A review of keratinocyte delivery to the wound bed. J Burn Care Rehabil. 2004 May-Jun;25(3):266-75. doi: 10.1097/01.bcr.0000124749.85552.cd. PMID 15273468
- [Result] Lumenta DB, Kamolz LP, Frey M. Adult burn patients with more than 60% TBSA involved-Meek and other techniques to overcome restricted skin harvest availability--the Viennese Concept. J Burn Care Res. 2009 Mar-Apr;30(2):231-42. doi: 10.1097/BCR.0b013e318198a2d6. PMID 19165111
- [Result] Svensjo T, Pomahac B, Yao F, Slama J, Wasif N, Eriksson E. Autologous skin transplantation: comparison of minced skin to other techniques. J Surg Res. 2002 Mar;103(1):19-29. doi: 10.1006/jsre.2001.6331. PMID 11855913
- [Result] Hackl F, Bergmann J, Granter SR, Koyama T, Kiwanuka E, Zuhaili B, Pomahac B, Caterson EJ, Junker JPE, Eriksson E. Epidermal regeneration by micrograft transplantation with immediate 100-fold expansion. Plast Reconstr Surg. 2012 Mar;129(3):443e-452e. doi: 10.1097/PRS.0b013e318241289c. PMID 22373992